CLINICAL TRIAL: NCT01233284
Title: A Phase II Randomised, Double-blind, Placebo Controlled, Cross-over Efficacy and Safety Comparison of Three Doses of Tiotropium Inhalation Solution Delivered Via Respimat Inhaler (1.25, 2.5 and 5.0 Mcg Once Daily) Versus Placebo in Patients With Moderate Persistent Asthma.
Brief Title: Randomised, Double- Blind, Cross-over Efficacy and Safety Comparison of Three Different Doses of Tiotropium Administered Once Daily Versus Placebo in Patients With Moderate Persistent Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.380; 2010-018471-26 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

ARMS (4):
- tiotropium low dose once daily (Experimental): once daily, delivered by the Respimat® inhaler
  Interventions: Drug: tiotropium bromide 1.25µg once daily
- tiotropium medium dose once daily (Experimental): once daily, delivered by the Respimat® inhaler
  Interventions: Drug: tiotropium bromide 2.5µg once daily
- tiotropium high dose once daily (Experimental): once daily, delivered by the Respimat® inhaler
  Interventions: Drug: tiotropium bromide high dose once daily
- Placebo once daily (Placebo Comparator): once daily, delivered by the Respimat® inhaler
  Interventions: Drug: Tiotropium matching Placebo once daily

INTERVENTIONS:
Drug: tiotropium bromide 2.5µg once daily — Efficacy and safety comparison of 3 doses of inhaled tiotropium (1.25µg, 2.5µg and 5µg) versus placebo
  Arms: tiotropium medium dose once daily
Drug: Tiotropium matching Placebo once daily — Efficacy and safety comparison of 3 doses of inhaled tiotropium (1.25µg, 2.5µg and 5µg) versus placebo
  Arms: Placebo once daily
Drug: tiotropium bromide high dose once daily — Efficacy and safety comparison of 3 doses of inhaled tiotropium (1.25µg, 2.5µg and 5µg) versus placebo
  Arms: tiotropium high dose once daily
Drug: tiotropium bromide 1.25µg once daily — IMP
  Arms: tiotropium low dose once daily

SUMMARY:
Rationale for the current trial is to evaluate the efficacy and safety of three doses (1.25 µg, 2.5 µg and 5.0 µg ex mouthpiece) of tiotropium inhalation solution in patients with moderate persistent asthma who are still symptomatic despite regular maintenance therapy with inhaled corticosteroids (ICS).

The data collected in the present trial will provide useful information to health care providers and patients regarding the efficacy and safety of a once daily inhalation of three different doses of tiotropium solution delivered by the Respimat® inhaler in addition to inhaled corticosteroids in the treatment of not fully controlled moderate asthma in comparison to placebo. The Pharmacokinetics (PK) of tiotropium is well established in COPD patients. However, there is currently no PK data available for the 3 doses of tiotropium being tested in this trial in patients with moderate persistent asthma. Tiotropium is a once daily drug. Hence, the rationale for blood and urine sampling for PK analysis over 24 hours in a subset of patients is to confirm the PK of the 3 doses in moderate asthma patients. Rationale for the 24-hour pulmonary function test sub-investigation is to demonstrate that a once daily dosing of tiotropium inhalation solution is effective and safe in the treatment of moderate persistent asthma.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign and date an Informed Consent Form consistent with the Harmonised Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local legislation prior to participation in the trial (i.e. prior to any trial procedures, including any pre-trial washout of medications and medication restrictions for pulmonary function test at Visit 1).
2. Male or female patients aged between 18 and 75 years (at date of informed consent).
3. All patients must have at least a 3 month history of asthma at the time of enrolment into the trial. The diagnosis should be confirmed at Visit 1 by fulfilling inclusion criterion no. 5.
4. The initial diagnosis of asthma must have been made before the patient's age of 40.
5. The diagnosis of asthma has to be confirmed at Visit 1 with a bronchodilator reversibility (15 to 30 minutes after 4 puffs of 100 µg salbutamol) resulting in a Forced Expiratory Volume in one second (FEV1) increase of = 12% and = 200mL.
6. All patients must have been on maintenance treatment with a medium, stable dose of inhaled corticosteroids (alone or in a fixed combination with a long acting or short acting beta agonist [LABA or SABA]) for at least 4 weeks prior to Visit 1.
7. All patients must be symptomatic at Visit 1 (screening) and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ) mean score of = 1.5.
8. All patients must have a pre-bronchodilator FEV1 = 60% and = 90% of predicted normal at Visit 1. Predicted normal values will be calculated according to the European Community for Steel and Coal (ECSC).
9. Variation of absolute FEV1 values of Visit 1 (pre-bronchodilator) as compared to Visit 2 (pre-dose) must be within ± 30%.
10. Patients must be never-smokers or ex-smokers who stopped smoking at least one year prior to enrolment (Visit 0) and who have a smoking history of less than 10 pack years.
11. Patients must be able to use the Respimat® inhaler correctly.
12. Patients must be able to perform all trial related procedures including technically acceptable pulmonary function tests and use of electronic diary/peak flow meter (diary compliance of at least 80% is required).

Exclusion criteria:

1. Patients with a significant disease other than asthma.
2. Patients with a clinically relevant abnormal screening (Visit 1) haematology or blood chemistry if the abnormality defines a significant disease as defined in exclusion criterion 1.
3. Patients with a recent history (i.e. six months or less) of myocardial infarction.
4. Patients who have been hospitalised for cardiac failure during the past year.
5. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year.
6. Patients with lung diseases other than asthma.
7. Patients with known active tuberculosis.
8. Patients with malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years.
9. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion no. 1.
10. Patients with known moderate to severe renal impairment.
11. Patients with known narrow angle glaucoma or any other disease where anticholinergic treatment is contraindicated.
12. Patients with significant symptomatic prostatic hyperplasia or bladder-neck obstruction. Patients whose symptoms are controlled on treatment may be included.
13. Patients with significant alcohol or drug abuse within the past two years (to the discretion of the investigator).
14. Patients who are currently in a pulmonary rehabilitation program or have completed pulmonary rehabilitation program in the 6 weeks prior to Visit 1 (screening) or who will start a rehabilitation program during the study.
15. Patients with known hypersensitivity to anticholinergic drugs, Benzalkonium chloride (BAC), Ethylenediaminetetraacetate (EDTA) or any other components of the study medication delivery system (Respimat®/ tiotropium inhalation solution).
16. Pregnant or nursing woman.
17. Women of childbearing potential not using a highly effective method of birth control.
18. Patients who have taken an investigational drug within four weeks prior to Visit 1.
19. Patients who have been treated with beta-blocker medication within four weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2). Topical cardio-selective beta-blocker eye medications for non-arrow angle glaucoma are allowed.
20. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva®) within four weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
21. Patients who have been treated with oral or patch beta-adrenergics within four weeks prior to Visit 1 and/or during the Screening period (period between Visit 1 and Visit 2)
22. Patients who have been treated with oral corticosteroids within four weeks prior to Visit 1 and/or during the screening period.
23. Patients who have been treated with anti-Immunoglobuline E (anti-IgE) antibodies, e.g. omalizumab, within 6 months prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
24. Patients who have been treated with cromone within two weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
25. Patients who have been treated with methylxanthines or phosphodiesterase 4 inhibitors within two weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
26. Patients who have been treated with other non-approved and according to international guidelines not recommended experimental drugs for routine asthma therapy (e.g. Tumor Necrosis Factor (TNF)-alpha blockers, methotrexate, cyclosporin) within four weeks prior to Visit 1 and/or during the screening period (period between Visit 1 and Visit 2).
27. Patient with any asthma exacerbation or respiratory tract infection in the 4 weeks prior to visit 1 and/or during the screening period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- Austria (5):
  - 205.380.43002 Boehringer Ingelheim Investigational Site, Hallein
  - 205.380.43004 Boehringer Ingelheim Investigational Site, Linz
  - 205.380.43005 Boehringer Ingelheim Investigational Site, Neumarkt am Wallersee
  - 205.380.43001 Boehringer Ingelheim Investigational Site, Schlüsslberg
  - 205.380.43003 Boehringer Ingelheim Investigational Site, Thalheim bei Wels
- Germany (9):
  - 205.380.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 205.380.49010 Boehringer Ingelheim Investigational Site, Berlin
  - 205.380.49003 Boehringer Ingelheim Investigational Site, Frankfurt
  - 205.380.49004 Boehringer Ingelheim Investigational Site, Hamburg
  - 205.380.49007 Boehringer Ingelheim Investigational Site, Hanover
  - 205.380.49009 Boehringer Ingelheim Investigational Site, Mainz
  - 205.380.49008 Boehringer Ingelheim Investigational Site, Schwerin
  - 205.380.49001 Boehringer Ingelheim Investigational Site, Wiesbaden
  - 205.380.49005 Boehringer Ingelheim Investigational Site, Wiesloch
- Ukraine (5):
  - 205.380.38005 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 205.380.38003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.380.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 205.380.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 205.380.38002 Boehringer Ingelheim Investigational Site, Kiev

REFERENCES:
- [Derived] Beeh KM, Moroni-Zentgraf P, Ablinger O, Hollaenderova Z, Unseld A, Engel M, Korn S. Tiotropium Respimat(R) in asthma: a double-blind, randomised, dose-ranging study in adult patients with moderate asthma. Respir Res. 2014 Jun 3;15(1):61. doi: 10.1186/1465-9921-15-61. PMID 24890738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 149 patients were randomised and treated, 141 patients completed the trial.
Pre-assignment Details: Randomised, double-blind, placebo controlled, cross-over design without washout phase between the four periods. Patients were randomized to one of the 4 sequences (ABCD, DCBA, BDAC, CADB). For one patient treatment 2 and treatment 3 were interchanged (resulting sequence DBCA).
Groups:
- Tio R5 Once Daily(qd)/Tio R1.25 qd/Placebo/Tio R2.5 qd: Patients treated with Tiotropium 5 mcg in period 1 (evening), with Tiotropium 1.25 mcg in period 2 (evening), with a matching Placebo in period 3 (evening) and with Tiotropium 2.5 mcg in period 4 (evening). All products were delivered by the Respimat inhaler as add-on therapy to inhaled corticosteroids (ICS). No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Tio R2.5 qd/Placebo/Tio R1.25 qd/Tio R5 qd: Patients treated with Tiotropium 2.5 mcg in period 1 (evening), with a matching Placebo in period 2 (evening), with Tiotropium 1.25 mcg in period 3 (evening) and with Tiotropium 5 mcg in period 4 (evening). All products were delivered by the Respimat inhaler as add-on therapy to ICS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Tio R1.25 qd/Tio R2.5 qd/Tio R5 qd/Placebo: Patients treated with Tiotropium 1.25 mcg in period 1 (evening), with Tiotropium 2.5 mcg in period 2 (evening), with Tiotropium 5 mcg in period 3 (evening) and with a matching placebo in period 4 (evening). All products were delivered by the Respimat inhaler as add-on therapy to inhaled corticosteroid ICS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Placebo/Tio R5 qd/Tio R2.5 qd/Tio R1.25 qd: Patients treated with a matching Placebo in period 1 (evening), with Tiotropium 5 mcg in period 2 (evening), with Tiotropium 2.5 mcg in period 3 (evening) and with Tiotropium 1.25 mcg in period 4 (evening). All products were delivered by the Respimat inhaler as add-on therapy to ICS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
- Placebo/Tio R2.5 qd/Tio R5 qd/Tio R1.25 qd: Patient treated with a matching Placebo in period 1 (evening), with Tiotropium 2.5 mcg in period 2 (evening), with Tiotropium 5 mcg in period 3 (evening) and with Tiotropium 1.25 mcg in period 4 (evening). All products were delivered by the Respimat inhaler as add-on therapy to ICS. No washouts (off-treatment periods) between treatments. Duration of each treatment period was 4 weeks.
Period: Period 1 (4 Weeks)
Arm/Group | Tio R5 Once Daily(qd)/Tio R1.25 qd/Placebo/Tio R2.5 qd | Tio R2.5 qd/Placebo/Tio R1.25 qd/Tio R5 qd | Tio R1.25 qd/Tio R2.5 qd/Tio R5 qd/Placebo | Placebo/Tio R5 qd/Tio R2.5 qd/Tio R1.25 qd | Placebo/Tio R2.5 qd/Tio R5 qd/Tio R1.25 qd
Started | 37 | 38 | 38 | 35 | 1
Completed | 36 | 37 | 37 | 35 | 1
Not Completed | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: Period 2 (4 Weeks)
Arm/Group | Tio R5 Once Daily(qd)/Tio R1.25 qd/Placebo/Tio R2.5 qd | Tio R2.5 qd/Placebo/Tio R1.25 qd/Tio R5 qd | Tio R1.25 qd/Tio R2.5 qd/Tio R5 qd/Placebo | Placebo/Tio R5 qd/Tio R2.5 qd/Tio R1.25 qd | Placebo/Tio R2.5 qd/Tio R5 qd/Tio R1.25 qd
Started | 36 | 37 | 37 | 35 | 1
Completed | 36 | 37 | 36 | 35 | 1
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Period 3 (4 Weeks)
Arm/Group | Tio R5 Once Daily(qd)/Tio R1.25 qd/Placebo/Tio R2.5 qd | Tio R2.5 qd/Placebo/Tio R1.25 qd/Tio R5 qd | Tio R1.25 qd/Tio R2.5 qd/Tio R5 qd/Placebo | Placebo/Tio R5 qd/Tio R2.5 qd/Tio R1.25 qd | Placebo/Tio R2.5 qd/Tio R5 qd/Tio R1.25 qd
Started | 36 | 37 | 36 | 35 | 1
Completed | 36 | 37 | 35 | 34 | 1
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0
Period: Period 4 (4 Weeks)
Arm/Group | Tio R5 Once Daily(qd)/Tio R1.25 qd/Placebo/Tio R2.5 qd | Tio R2.5 qd/Placebo/Tio R1.25 qd/Tio R5 qd | Tio R1.25 qd/Tio R2.5 qd/Tio R5 qd/Placebo | Placebo/Tio R5 qd/Tio R2.5 qd/Tio R1.25 qd | Placebo/Tio R2.5 qd/Tio R5 qd/Tio R1.25 qd
Started | 36 | 37 | 35 | 34 | 1
Completed | 36 | 36 | 35 | 33 | 1
Not Completed | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Total: Total number of patients randomised and treated in the study.
Arm/Group | Baseline Total
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 67

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Peak Within 0-3 Hours Post-dose Response
Description: Mixed model repeated measurement (MMRM) results. Response was defined as change from baseline at the end of of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 10 minutes (min) before drug administration and 30 min, 1h, 2h, 3h after drug administration
Population: Full analysis set (FAS) reduced to patients with non-missing FEV1 data. The FAS is defined as patients randomised, treated, with baseline data and at least one on-treatment efficacy measurement after 4 weeks on treatment within a period.
Measure: Mean (Standard Error); unit: Litre
Groups:
- Placebo: Matching Placebo qd in the evening delivered by the Respimat inhaler.
- Tio R1.25 qd: Tiotropium 1.25 mcg qd in the evening delivered by the Respimat inhaler as add-on therapy to ICS.
- Tio R2.5 qd: Tiotropium 2.5 mcg qd in the evening delivered by the Respimat inhaler as add-on therapy to ICS.
- Tio R5 qd: Tiotropium 5 mcg qd in the evening delivered by the Respimat inhaler as add-on therapy to ICS.
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre | 0.116 (0.027) | 0.255 (0.027) | 0.244 (0.027) | 0.304 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.138, 95% CI [0.090 to 0.186], Standard Error of Mean 0.024 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.128, 95% CI [0.080 to 0.176], Standard Error of Mean 0.024 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.188, 95% CI [0.140 to 0.236], Standard Error of Mean 0.024 — Tio R5 qd minus Placebo

2. Secondary Outcome: Trough FEV1 Response
Description: MMRM results. Response was defined as change from baseline at the end of of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. Trough FEV1 was measured just prior to the last administration of randomised treatment.
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing FEV1 data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre | 0.006 (0.027) | 0.131 (0.027) | 0.138 (0.027) | 0.149 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.125, 95% CI [0.078 to 0.173], Standard Error of Mean 0.024 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.132, 95% CI [0.084 to 0.179], Standard Error of Mean 0.024 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.143, 95% CI [0.096 to 0.191], Standard Error of Mean 0.024 — Tio R5 qd minus Placebo

3. Secondary Outcome: FEV1 Area Under the Curve 0-3 Hours (AUC0-3h) Response
Description: MMRM results. Response was defined as change from baseline at the end of of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC0-3h was calculated using the trapezoidal rule divided by the observation time (3 hours) to report in litres.
Time Frame: 10 minutes (min) before drug administration and 30 min, 1h, 2h, 3h after drug administration
Population: FAS reduced to patients with non-missing FEV1 data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre | 0.025 (0.027) | 0.154 (0.027) | 0.152 (0.027) | 0.203 (0.027)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.129, 95% CI [0.083 to 0.175], Standard Error of Mean 0.023 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.127, 95% CI [0.081 to 0.172], Standard Error of Mean 0.023 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.178, 95% CI [0.132 to 0.224], Standard Error of Mean 0.023 — Tio R5 qd minus Placebo

4. Secondary Outcome: Forced Vital Capacity (FVC) Peak Within 0-3 Hours Post-dose Response
Description: MMRM results. Response was defined as change from baseline at the end of of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: 10 minutes (min) before drug administration and 30 min, 1h, 2h, 3h after drug administration
Population: FAS reduced to patients with non-missing FVC data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre | 0.092 (0.034) | 0.171 (0.034) | 0.163 (0.034) | 0.229 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.079, 95% CI [0.026 to 0.132], Standard Error of Mean 0.027 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.0087, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.071, 95% CI [0.018 to 0.124], Standard Error of Mean 0.027 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.137, 95% CI [0.085 to 0.190], Standard Error of Mean 0.027 — Tio R5 qd minus Placebo

5. Secondary Outcome: Trough FVC Response
Description: MMRM results. Response was defined as change from baseline at the end of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. Trough FVC was measured just prior to the last administration of randomised treatment.
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing FVC data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre | 0.004 (0.035) | 0.058 (0.035) | 0.076 (0.035) | 0.102 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.0732, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.054, 95% CI [-0.005 to 0.113], Standard Error of Mean 0.030 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.0177, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.072, 95% CI [0.012 to 0.131], Standard Error of Mean 0.030 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.098, 95% CI [0.039 to 0.157], Standard Error of Mean 0.030 — Tio R5 qd minus Placebo

6. Secondary Outcome: FVC AUC0-3h Response
Description: MMRM results. Response was defined as change from baseline at the end of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. FVC AUC0-3h was calculated using the trapezoidal rule divided by the observation time (3 hours) to report in litres.
Time Frame: 10 minutes (min) before drug administration and 30 min, 1h, 2h, 3h after drug administration
Population: FAS reduced to patients with non-missing FVC data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre | -0.028 (0.034) | 0.036 (0.034) | 0.047 (0.034) | 0.110 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.0149, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.064, 95% CI [0.013 to 0.115], Standard Error of Mean 0.026 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.0043, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.075, 95% CI [0.024 to 0.126], Standard Error of Mean 0.026 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.138, 95% CI [0.086 to 0.189], Standard Error of Mean 0.026 — Tio R5 qd minus Placebo

7. Secondary Outcome: Individual FEV1 Over Time (at Each Timepoint at Visits) Response
Description: MMRM results. Response was defined as change from baseline at the end of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline.
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing FEV1 data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre
  Timepoint -0:10 | 0.006 (0.027) | 0.131 (0.027) | 0.138 (0.027) | 0.149 (0.027)
  Timepoint 0:30 | 0.029 (0.028) | 0.160 (0.028) | 0.163 (0.028) | 0.209 (0.028)
  Timepoint 1:00 | 0.026 (0.029) | 0.148 (0.029) | 0.156 (0.029) | 0.205 (0.029)
  Timepoint 2:00 | 0.033 (0.029) | 0.158 (0.029) | 0.149 (0.029) | 0.218 (0.029)
  Timepoint 3:00 | 0.013 (0.029) | 0.160 (0.029) | 0.148 (0.029) | 0.191 (0.029)

8. Secondary Outcome: Individual FVC Over Time (at Each Timepoint at Visits) Response
Description: as for outcome 7
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing FVC data.
Measure: Mean (Standard Error); unit: Litre
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre
  Timepoint -0:10 | 0.004 (0.035) | 0.058 (0.035) | 0.076 (0.035) | 0.102 (0.035)
  Timepoint 0:30 | -0.028 (0.035) | 0.042 (0.035) | 0.060 (0.035) | 0.124 (0.035)
  Timepoint 1:00 | -0.031 (0.036) | 0.024 (0.036) | 0.041 (0.036) | 0.112 (0.036)
  Timepoint 2:00 | -0.022 (0.036) | 0.037 (0.036) | 0.045 (0.036) | 0.119 (0.036)
  Timepoint 3:00 | -0.050 (0.036) | 0.036 (0.036) | 0.033 (0.036) | 0.078 (0.036)

9. Secondary Outcome: Individual Peak Expiratory Flow (PEF) Over Time (at Each Timepoint at Visits) Response
Description: as for outcome 7
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing PEF data.
Measure: Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 144 | 144 | 144 | 143
Litre/min
  Timepoint -0:10 | 11.038 (4.804) | 30.567 (4.802) | 33.903 (4.804) | 34.787 (4.812)
  Timepoint 0:30 | 8.235 (4.949) | 32.163 (4.947) | 37.149 (4.949) | 39.325 (4.957)
  Timepoint 1:00 | 6.095 (5.074) | 34.070 (5.072) | 36.851 (5.074) | 41.260 (5.082)
  Timepoint 2:00 | 7.237 (5.039) | 34.544 (5.037) | 36.972 (5.039) | 42.694 (5.047)
  Timepoint 3:00 | 5.046 (5.024) | 34.620 (5.022) | 37.283 (5.024) | 40.624 (5.033)

10. Secondary Outcome: Mean Pre-dose Morning PEF (PEF a.m.) Response During the Last Week on Treatment
Description: MMRM results. Response was defined as change from baseline at the end of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. Weekly means obtained during the last week of each period of randomised treatment will be compared (measured by patients at home using the AM2+ device).
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing morning PEF data.
Measure: Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Litre/min | 4.395 (4.573) | 22.944 (4.543) | 22.290 (4.543) | 25.241 (4.559)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 18.550, 95% CI [11.204 to 25.895], Standard Error of Mean 3.737 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 17.895, 95% CI [10.550 to 25.240], Standard Error of Mean 3.737 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 20.846, 95% CI [13.497 to 28.195], Standard Error of Mean 3.739 — Tio R5 qd minus Placebo

11. Secondary Outcome: Mean Pre-dose Evening PEF (PEF p.m.) Response During the Last Week on Treatment
Description: as for outcome 10
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing evening PEF data.
Measure: Mean (Standard Error); unit: Litre/min
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Litre/min | 3.833 (4.363) | 25.084 (4.331) | 18.410 (4.331) | 25.414 (4.348)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 21.251, 95% CI [13.840 to 28.662], Standard Error of Mean 3.770 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 14.577, 95% CI [7.166 to 21.988], Standard Error of Mean 3.770 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 21.581, 95% CI [14.166 to 28.997], Standard Error of Mean 3.773 — Tio R5 qd minus Placebo

12. Secondary Outcome: PEF Variability Response (Last Week on Treatment)
Description: MMRM results. Response was defined as change from baseline at the end of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. PEF variability is the absolute difference between morning and evening PEF value divided by the mean of these two values, expressed as a percent . Weekly means obtained during the last week of each period of randomised treatment will be compared.
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing morning and evening PEF data.
Measure: Mean (Standard Error); unit: Percentage of the mean daily PEF
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Percentage of the mean daily PEF | -0.171 (0.615) | -0.285 (0.609) | -0.711 (0.609) | -0.248 (0.612)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.8574, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.114, 95% CI [-1.363 to 1.134], Standard Error of Mean 0.635 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.3954, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.540, 95% CI [-1.789 to 0.708], Standard Error of Mean 0.635 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.9034, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.077, 95% CI [-1.327 to 1.173], Standard Error of Mean 0.636 — Tio R5 qd minus Placebo

13. Secondary Outcome: Mean Number of Puffs of Rescue Medication During the Whole Day (Last Week on Treatment, Response Values)
Description: as for outcome 10
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing data for rescue medication.
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Puffs | -0.569 (0.122) | -0.802 (0.121) | -0.783 (0.121) | -0.769 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.0296, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.233, 95% CI [-0.443 to -0.023], Standard Error of Mean 0.107 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.0454, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.214, 95% CI [-0.424 to -0.004], Standard Error of Mean 0.107 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0610, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.201, 95% CI [-0.410 to 0.009], Standard Error of Mean 0.107 — Tio R5 qd minus Placebo

14. Secondary Outcome: Mean Number of Puffs of Rescue Medication During Daytime (Last Week on Treatment, Response Values)
Description: as for outcome 10
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing data for rescue medication.
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Puffs | -0.314 (0.071) | -0.463 (0.071) | -0.452 (0.071) | -0.425 (0.071)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.0183, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.149, 95% CI [-0.273 to -0.025], Standard Error of Mean 0.063 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.0288, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.138, 95% CI [-0.262 to -0.014], Standard Error of Mean 0.063 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.0781, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.111, 95% CI [-0.235 to 0.013], Standard Error of Mean 0.063 — Tio R5 qd minus Placebo

15. Secondary Outcome: Mean Number of Puffs of Rescue Medication During Nighttime (Last Week on Treatment, Response Values)
Description: as for outcome 10
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing data for rescue medication.
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Puffs | -0.273 (0.064) | -0.357 (0.063) | -0.341 (0.063) | -0.360 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.1303, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.084, 95% CI [-0.193 to 0.025], Standard Error of Mean 0.055 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.2191, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.068, 95% CI [-0.177 to 0.041], Standard Error of Mean 0.055 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.1163, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.087, 95% CI [-0.196 to 0.022], Standard Error of Mean 0.056 — Tio R5 qd minus Placebo

16. Secondary Outcome: Mean Number of Night Awakenings During the Last Week on Treatment (Score, Response Values)
Description: as for outcome 10
Time Frame: Baseline and 4 weeks
Population: FAS reduced to patients with non-missing data for nighttime awakenings
Measure: Mean (Standard Error); unit: Night awakenings
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 142 | 146 | 146 | 144
Night awakenings | -0.156 (0.034) | -0.166 (0.034) | -0.162 (0.034) | -0.187 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Test type: Superiority or Other; p = 0.7501, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.010, 95% CI [-0.073 to 0.052], Standard Error of Mean 0.032 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Test type: Superiority or Other; p = 0.8401, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.006, 95% CI [-0.069 to 0.056], Standard Error of Mean 0.032 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Test type: Superiority or Other; p = 0.3237, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = -0.031, 95% CI [-0.094 to 0.031], Standard Error of Mean 0.032 — Tio R5 qd minus Placebo

17. Secondary Outcome: FEV1 Area Under the Curve Within 24 Hours (h) Response (FEV1 AUC0-12h, FEV1 AUC12-24h, FEV1 AUC0-24h)
Description: MMRM results. Response was defined as change from baseline at the end of of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. FEV1 AUC0-12, FEV1 AUC12-24 and FEV1 AUC0-24 were calculated using the trapezoidal rule divided by the observation time (12h resp. 24h) to report in litres.
Time Frame: 10 minutes (min) before drug administration and 30 min, 1h, 2h, 3h, 4h, 11h 50min, 12h 30min, 13h, 14h, 15h, 16h, 18h, 20h, 22h, 23h, 23h 50min after drug administration
Population: FAS24 was defined as all patients in the FAS who gave informed consent for the 24-h PFT and who participated in this optional PFT.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 21 | 24 | 24 | 24
Litres
  FEV1 AUC0-12h | -0.013 (0.058) | 0.105 (0.055) | 0.134 (0.054) | 0.128 (0.054)
  FEV1 AUC12-24h | 0.012 (0.061) | 0.093 (0.058) | 0.148 (0.058) | 0.208 (0.057)
  FEV1 AUC0-24h | -0.001 (0.057) | 0.099 (0.054) | 0.141 (0.054) | 0.168 (0.053)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Comparison vs. Placebo for AUC0-12h; Test type: Superiority or Other; p = 0.1402, Mixed Models Analysis — MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [-0.040 to 0.276], Standard Error of Mean 0.079 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Comparison vs. Placebo for AUC0-12h; Test type: Superiority or Other; p = 0.0656, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.148, 95% CI 2-sided [-0.010 to 0.305], Standard Error of Mean 0.079 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Comparison vs. Placebo for AUC0-12h; Test type: Superiority or Other; p = 0.0766, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [-0.015 to 0.299], Standard Error of Mean 0.079 — Tio R5 qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Tio R1.25 qd; Comparison vs. Placebo for AUC12-24h; Test type: Superiority or Other; p = 0.3371, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.081, 95% CI 2-sided [-0.086 to 0.249], Standard Error of Mean 0.084 — Tio R1.25 qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Tio R2.5 qd; Comparison vs. Placebo for AUC12-24h; Test type: Superiority or Other; p = 0.1097, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.136, 95% CI 2-sided [-0.031 to 0.303], Standard Error of Mean 0.084 — Tio R2.5 qd minus Placebo
Statistical Analysis 6: Comparison: Placebo vs Tio R5 qd; Comparison vs. Placebo for AUC12-24h; Test type: Superiority or Other; p = 0.0220, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.196, 95% CI 2-sided [0.029 to 0.363], Standard Error of Mean 0.084 — Tio R5 qd minus Placebo
Statistical Analysis 7: Comparison: Placebo vs Tio R1.25 qd; Comparison vs. Placebo for AUC0-24h; Test type: Superiority or Other; p = 0.2062, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.100, 95% CI 2-sided [-0.056 to 0.256], Standard Error of Mean 0.078 — Tio R1.25 qd minus Placebo
Statistical Analysis 8: Comparison: Placebo vs Tio R2.5 qd; Comparison vs. Placebo for AUC0-24h; Test type: Superiority or Other; p = 0.0731, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [-0.014 to 0.297], Standard Error of Mean 0.078 — Tio R2.5 qd minus Placebo
Statistical Analysis 9: Comparison: Placebo vs Tio R5 qd; Comparison vs. Placebo for AUC0-24h; Test type: Superiority or Other; p = 0.0333, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.169, 95% CI 2-sided [0.014 to 0.324], Standard Error of Mean 0.078 — Tio R5 qd minus Placebo

18. Secondary Outcome: FVC Area Under the Curve Within 24 Hours (h) Response (FVC AUC0-12h, FVC AUC12-24h, FVC AUC0-24h)
Description: MMRM results. Response was defined as change from baseline at the end of of each 4-week treatment period. Means are adjusted for treatment, period, patient and study baseline. FVC AUC0-12, FVC AUC12-24 and FVC AUC0-24 were calculated using the trapezoidal rule divided by the observation time (12h resp. 24h) to report in litres.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Number analyzed (Participants) | 21 | 24 | 24 | 24
Litres
  FVC AUC0-12h | -0.052 (0.072) | 0.064 (0.068) | 0.157 (0.068) | 0.115 (0.068)
  FVC AUC12-24h | -0.021 (0.076) | 0.046 (0.071) | 0.177 (0.071) | 0.160 (0.071)
  FVC AUC0-24h | -0.036 (0.072) | 0.055 (0.067) | 0.167 (0.067) | 0.137 (0.067)
Statistical Analysis 1: Comparison: Placebo vs Tio R1.25 qd; Comparison vs. Placebo for AUC0-12h; Test type: Superiority or Other; p = 0.2451, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.116, 95% CI 2-sided [-0.081 to 0.312], Standard Error of Mean 0.099 — Tio R1.25 qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Tio R2.5 qd; Comparison vs. Placebo for AUC0-12h; Test type: Superiority or Other; p = 0.0379, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.209, 95% CI 2-sided [0.012 to 0.405], Standard Error of Mean 0.099 — Tio R2.5 qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio R5 qd; Comparison vs. Placebo for AUC0-12h; Test type: Superiority or Other; p = 0.0957, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.167, 95% CI 2-sided [-0.030 to 0.363], Standard Error of Mean 0.099 — Tio R5 qd minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Tio R1.25 qd; Comparison vs. Placebo for AUC12-24h; Test type: Superiority or Other; p = 0.5207, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.067, 95% CI 2-sided [-0.139 to 0.273], Standard Error of Mean 0.104 — Tio R1.25 qd minus Placebo
Statistical Analysis 5: Comparison: Placebo vs Tio R2.5 qd; Comparison vs. Placebo for AUC12-24h; Test type: Superiority or Other; p = 0.0606, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.198, 95% CI 2-sided [-0.009 to 0.404], Standard Error of Mean 0.104 — Tio R2.5 qd minus Placebo
Statistical Analysis 6: Comparison: Placebo vs Tio R5 qd; Comparison vs. Placebo for AUC12-24h; Test type: Superiority or Other; p = 0.0855, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.181, 95% CI 2-sided [-0.026 to 0.387], Standard Error of Mean 0.104 — Tio R5 qd minus Placebo
Statistical Analysis 7: Comparison: Placebo vs Tio R1.25 qd; Comparison vs. Placebo for AUC0-24h; Test type: Superiority or Other; p = 0.3564, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [-0.104 to 0.287], Standard Error of Mean 0.099 — Tio R1.25 qd minus Placebo
Statistical Analysis 8: Comparison: Placebo vs Tio R2.5 qd; Comparison vs. Placebo for AUC0-24h; Test type: Superiority or Other; p = 0.0424, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.203, 95% CI 2-sided [0.007 to 0.399], Standard Error of Mean 0.099 — Tio R2.5 qd minus Placebo
Statistical Analysis 9: Comparison: Placebo vs Tio R5 qd; Comparison vs. Placebo for AUC0-24h; Test type: Superiority or Other; p = 0.0815, Mixed Models Analysis; MMRM, adjusted for treatment, period, patient and study baseline; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [-0.022 to 0.370], Standard Error of Mean 0.099 — Tio R5 qd minus Placebo

ADVERSE EVENTS:
Time Frame: 4 weeks + 30 days if in last period
Arm/Group | Placebo | Tio R1.25 qd | Tio R2.5 qd | Tio R5 qd
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/146 | 0/147 | 2/146
Other Adverse Events (participants affected / at risk) | 0/144 | 0/146 | 0/147 | 0/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=144) | Tio R1.25 qd (N=146) | Tio R2.5 qd (N=147) | Tio R5 qd (N=146)
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.